CLINICAL TRIAL: NCT06337513
Title: Spondyloarthritis Inception Cohort of Southern Denmark
Acronym: SPINCODE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Danish Center for Expertise in Rheumatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SPINCODE (S-20230055)
Record Dates: First submitted 2024-03-12; First posted 2024-03-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Axial Spondyloarthritis; Back Pain
MeSH Terms: conditions — Axial Spondyloarthritis; Back Pain

STUDY DESIGN:
Intervention Model Description: In the rehabilitation feasibility study: pre-post design. In the rehabilitation RCT, participants are allocated to either the intervention or control group with standard care.
Who Masked: Outcomes Assessor
Masking Description: Blinding of the the health care professionals and patients is not possible in the rehabilitation intervention. The person analysing the data will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention consists of a physiotherapist-coordinated (PT) interdisciplinary outpatient rehabilitation for 6-months.
  Interventions: Other: Rehabilitation intervention
- Usual care (control group) (Active Comparator): Both groups are offered standard care.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Rehabilitation intervention — The intervention consists of a physiotherapist-coordinated (PT) interdisciplinary outpatient rehabilitation offer for 6-months.
  The intervention encompasses 3 individual sessions with the PT, if needed individual sessions with the interdisciplinary team (PT, occupational therapist, OT, nurse, and social worker) (a maximum of 6 hours), and patient education in two group seminars.
  Arms: Intervention group
Other: Usual care — Both the intervention and the control group will receive usual care.
  Arms: Usual care (control group)

SUMMARY:
People with axial spondyloarthritis (axSpA) experience a diagnostic delay of 6.5 years in men and up to 8.8 years in women. One of the reasons for the diagnostic delay seems to be limited awareness of the disease characteristics in the referring health care professionals in primary care. By raising awareness about the disease, the study aims at reducing the diagnostic delay and improving early treatment. In addition to diagnostic and pharmacological treatment, physical exercise and rehabilitation are recommended in people with axSpA. In Denmark, people with axSpA are only offered free of charge physiotherapy when the disease has progressed to a stage with radiographic changes of the spine even though people in the early stage of axSpA report a similar disease burden.

The overall objective of Spondyloarthritis Inception Cohort of Southern Denmark (SPINCODE) is to set up an axSpA inception cohort among individuals with low back pain ≥ 3 months who are considered to be at risk for axSpA. The investigators aim to learn more about the course of axSpA during the early stage of disease appropriately assess outcomes, including novel imaging techniques and identify predictive outcomes. Moreover, the investigators want to test the effect of an outpatient physiotherapist-coordinated rehabilitation intervention in people suspected of having axSpA.

DETAILED DESCRIPTION:
Spondyloarthritis (SpA) affects 0.1-3% of the population in Denmark, i.e. approximately 100.000 individuals. SpA encompasses among other diseases axial spondyloarthritis (axSpA). There is a diagnostic delay of 6.5 years in men and up to 8.8 years in women in people with axSpA and it may partly be due to a lack of awareness of possible SpA in the primary care sector. Structured exercise is recommended for people with axSpA by international organisations. Therefore, information about exercise safety and physical activity guidance by physiotherapists (PT) are recommended. At present, most people with axSpA are not offered support from PTs or occupational therapists in rheumatology outpatient clinics in Denmark, and not all see an outpatient rheumatology nurse for patient education and self-management support although this is recommended. The importance of coherence in rehabilitation across all levels in the health care system has been highlighted by the World Health Organisation (WHO). To gain and maintain benefits from the interdisciplinary rehabilitative initiatives in the rheumatology clinics, patients with axSpA need support in the transition from the rheumatology outpatient clinic to primary care to ensure long-term rehabilitation benefits. In summary, early referral and early rehabilitation in people with SpA are inadequate and need improvement.

Aims:

To set up an axSpA inception cohort among individuals with low back pain ≥ 3 months in the counties of Southern Jutland who are considered to be at risk for axSpA.

To describe the epidemiology, demographics, clinical, laboratory and imaging signatures in a population with low back pain suspected of axSpA and improve awareness about incipient axSpA.

To test the feasibility of a novel outpatient interdisciplinary rehabilitation intervention for patients with low back pain suspected of SpA

To evaluate and compare the effect of a novel outpatient interdisciplinary rehabilitation intervention (adjunct to pharmacological therapy) for patients with suspected SpA by studying differences in pain, fatigue, mental and physical functioning, work ability, physical activity levels and quality of life among those with and without a definite axSpA diagnosis

Methods:

The study consists of a medical part and a rehabilitation part. The medical part is planned as a prospective observational single centre cohort study of consecutive patients with low back pain ≥3 months and ≤ 3 years, symptom onset at age 18-45 years and suspected of axSpA, referred from the Counties of Southern Jutland, and followed at Danish Hospital for Rheumatic Diseases (DHR) for a consecutive period of two years. In order to diagnose axSpA and to improve diagnostic accuracy there will be used novel imaging techniques like low-dose computed tomography (ld-CT) and dual energy computed tomography (DECT) in addition to standard of care magnetic resonance imaging (MRI) of the sacroiliac joints (SIJ) and spine.

The rehabilitation design is developed in accordance with the Medical Research Council's framework for developing complex interventions. The design will be tested in a feasibility study, adapted as needed and planned to be tested in randomised controlled study (RCT) in addition to pharmacological treatment.

SPINCODE is overall a two-year observational cohort study. The rehabilitation study is a 6-months intervention study followed by a 18-months observational follow-up study. The rehabilitation feasibility study will be a pre-post design without a control group, the design is expected to be adapted and tested in a RCT study.

The intervention consists of a physiotherapist-coordinated (PT) interdisciplinary outpatient rehabilitation offer for 6-months. The intervention encompasses 3 individual sessions with the PT, if needed individual consultations from the interdisciplinary team (PT, occupational therapist, OT, nurse, and social worker) (a maximum of 6 hours), and patient education in two group seminars.The individual sessions are based on the following theories: self-efficacy, Focused and Acceptance Commitment Therapy (FACT), and shared decision making/person-centered care. Overall, the PT offers advise on physical activity and supports the patient's self-management. The counselling is person-centered and derived from the shared goal setting at the initial assessment. The PT has a coordinating role both internal by referring the patient to other health care professionals from the interdisciplinary team if needed and an external by supporting the patient in finding and take actions on relevant offers in the municipality. Moreover, if a patient has a private PT, the patient's PT is offered an online support from the coordinating PT. The group sessions are two 2-hour group sessions with patient education delivered by the interdisciplinary team (PT, rheumatologist, OT, social worker, and nurse). Moreover, it is an opportunity for peer support.

Study setting:

SPINCODE will be carried out at the Danish Hospital for Rheumatic Diseases, located in the city of Sønderborg, Denmark.

Recruitment:

Patients with low back pain suspected of axSpA will be referred according to the referral algorithm by: general practitioners (GPs), ophthalmologists and dermatologists from the Counties of Southern Jutland, departments of ophthalmology and gastroenterology at the Hospital of Southern Jutland, University Hospital of Southern Denmark.

Referring physicians will inform patients about the project prior to the referral to the DHR and note in the referral whether the patient has given permission to receive an introduction call from the research nurse. If this permission is not noted in the referral, first contact will be established at the first meeting in the outpatient clinic.

Consultants responsible for visitation of referrals to the DHR will be prepared to screen referrals for patients with suspected axSpA according to the inclusion and exclusion criteria during the study period.

If the patient has been introduced to the project and asked permission to receive information as described above, the research nurse will call the patient, inform about the study and perform a pre-screening to ensure that patients meeting to the screening visit most likely also can be included into the study. Furthermore, the research nurse will ask permission to send written information, patients' rights and the consent form electronically to the patient's electronic mail box to ensure a consideration period of at least seven days.

The trial participants are offered verbal information upon physical attendance. If trial participants do not want oral information when physically present, the right to a bystander is ensured, by agreement on a telephone appointment, when participation of a bystander during the telephone conversation can be realized.

Randomisation and blinding:

If the rehabilitation feasibility study's findings are promising, the rehabilitation study will afterwards be tested in a randomised controlled study with a 1:1 allocation to either an outpatient physiotherapist-coordinated interdisciplinary rehabilitation (in addition to pharmacological treatment) or standard care.

Due to the nature of the rehabilitation intervention, it is not possible to blind the healthcare professionals and the patients. The statistical analyses will be performed blinded to group allocation.

Data collection:

Outcomes in SPINCODE will be tested at baseline/visit 1 (0-6 weeks), visit 3 (6 months), visit 4 (1 year), visit 5 (1½ year), and visit 6 (2 years).

Ethics:

The participants will be informed verbally and in writing about the study before providing their written consent to participate before the first consultation. The study will be conducted in accordance with the Helsinki Declaration. The leaflet," Research subjects' rights in health science research" published by the Danish National Committee on Health Research Ethics, is provided to all participants. The Regional Committees on Health Research Ethics has approved the study (Project ID S-20230055). Data will be stored and managed in the Open Patient Data Explorative Network (OPEN), which adheres to the European General Data Protection Regulations and the Danish data protection law.

ELIGIBILITY:
Patients with low back pain suspected of axSpA will be included based on the following inclusion and exclusion criteria.

Inclusion Criteria:

* Age ≥ 18 years
* Age at symptom onset ≤ 45 years
* Currently diagnosed with undifferentiated lower back pain
* Onset of back pain ≥ 3 months ≤ 3 years at referral
* Diagnosed with anterior uveitis (AU) and/or psoriasis and/or inflammatory bowel disease (IBD) regardless of human leukocyte antigen B27 (HLA-B27) status
* HLA-B 27 positivity (obligatory in case of absence of AU, psoriasis or IBD)
* Imaging findings suggestive of axSpA as defined by trained musculoskeletal radiologists, regardless of HLA-B27 status
* Patients capable of giving written informed consent

Exclusion Criteria:

* Age < 18 years
* Age at symptom onset > 45 years
* Recurrent episodes of low back pain for >3 years
* Incapable of complying with the examination program for physical or mental reasons
* Not able to provide written consent
* Not able to understand Danish
* A priori SpA diagnosis
* Contradictions to MRI
* Treatment with disease modifying antirheumatic drugs (DMARDs) for other conditions
* Pregnancy

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Clinicians diagnosis of axSpA | Baseline, week 6, 24, 48, 72 and 96
  The treating rheumatologists diagnosis of axial spondyloarthritis
Health related quality of life | Baseline, week 6, week 24, 48, 72 and 96
  EuroQol -5-dimension 5 level-version (EQ-5D-5L) is a generic measure to assess population health. Includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The EQ-5D-5L index ranges from 0.00 to 1.00. The highest score, the better health related quality of life

SECONDARY OUTCOMES:
axSpA disease activity | Baseline, week 24, 48, 72 and 96
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). The scale ranges from 0-100. The higher number, the more active disease.
axSpA disease mobility | Baseline, week 6, 24, 48 and 96
  Bath Ankylosing Spondylitis Metrology Index (BASMI).The scale ranges from 0-100. The higher number, the more impaired mobility.
axSpA patient-reported physical function | Baseline, week 24, 48, 72 and 96
  Bath Ankylosing Spondylitis Functional Index (BASFI). The scale ranges from 0-100. The higher number, the more impaired physical function.
Inflammatory back pain (IBP) symptoms | Baseline, week 6, 12, 24, 48, 72, 96
  Symptoms characteristic for inflammatory back pain
Physical examination I | Baseline, week 6, 24, 48, 72 and 96
  swollen joint count (SIJC)/tender joint count (TJC) - 46 joints will be assessed for tenderness and 44 joints will be assessed for swollenness (yes or no)
Physical examination II | Baseline, week 6, 24, 48, 72 and 96
  Enthesitis will be assessed according to the Spondyloarthritis Research Consortium of Canada score for enthesitis (SPARCC score), which ranges from 0-16. The higher the score, the more enthesitis.
Symptomatic SpA features I | Baseline, week 6, 24, 48, 72 and 96
  Elevated C-reactive protein (CRP) due to disease activity, measured in milligram per liter
Symptomatic SpA features II | Baseline, week 6, 24, 48, 72 and 96
  presence of psoriasis at skin and nails
Symptomatic SpA features III | Baseline, week 6, 24, 48, 72 and 96
  presence of anterior uveitis
Symptomatic SpA features IV | Baseline, week 6, 24, 48, 72 and 96
  presence of inflammatory bowel disease
Symptomatic SpA features V | Baseline, week 6, 24, 48, 72 and 96
  presence of dactylitis
Symptomatic SpA features VI | Baseline, week 6, 24, 48, 72 and 96
  presence of heel enthesitis
Physicians global assessment of disease activity | Baseline, week 6, 24, 48, 72 and 96
  The treating physicians overall assessment of disease activity on a visual analog scale (VAS 0-10). The higher number, the more active disease.
Magnetic resonance imaging of sacroiliac joints (SIJ) and spine | Baseline and week 96
  the radiologists confidence in diagnosis of axSpA will be recorded on a numeric scale ranging from -5 (definitely not axSpA) to +5 (definitely axSpA)
low dose computed tomography of SIJ and spine | Baseline and week 96
  the radiologists confidence in diagnosis of axSpA will be recorded on a numeric scale ranging from -5 (definitely not axSpA) to +5 (definitely axSpA)
dual energy computed tomography of SIJ | Baseline and week 96
  the radiologists confidence in diagnosis of axSpA will be recorded on a numeric scale ranging from -5 (definitely not axSpA) to +5 (definitely axSpA)
radiography SIJ | Baseline
  the radiologist will assess fulfillment of modified New York criteria (yes or no)
Work | Week 6, 24, 48, 72 and 96
  Work Productivity and Activity Impairment questionnaire, general health (WPAI:GH). The result is presented in percentages. The higher number, the worse work ability.
Fatigue | Week 6, 24, 48, 72 and 96
  Bristol Rheumatoid Arthritis Fatigue Numeric Rating Scale (BRAF-NRS). There are 3 NRS scales investigating severity, impact and coping regarding fatigue. The scales ranges from 0-10. The higher number, the more fatigued.
Physical activity | Week 6, 24, 48, 72 and 96
  Physical Activity Scale version2 (PAS2). PAS2 is expressed in minutes and measures both sedentary time and time being physically active.
Sleep | Week 6, 24, 48, 72 and 96
  Insomnia Severity Index (ISI). The scale ranges from 0-28. The higher number, the more impaired sleep.
Self-efficacy | Week 6, 24, 48, 72 and 96
  Self-Efficacy for Managing Chronic Diseases 6-item Scale (SES6G). The scale ranges from 1-10. The higher number, the higher degree of self-efficacy.
Objective physical function | Week 6, 24, 48, 72 and 96
  Ankylosing spondylitis performance index (ASPI). The performance is measured in seconds and a faster time means a better physical function.
Aerobic capacity | Week 6, 24, 48, 72 and 96
  Indirect maximal aerobic capacity testing (modified Balke protocol)

OTHER OUTCOMES:
Patient global assessment | Baseline, week 24, 48, 72 and 96
  Patient global assessment of health status (VAS 0-10)
Acceptable state | Week 6, 24, 48, 72 and 96
  Patient acceptable symptom state (PASS)
Mental state | Week 6, 24, 48, 72 and 96
  Anxiety and depression questions. The scale ranges from 0-3. The higher number, the more anxious or depressed.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Kroeber, MD, Principal Investigator — Danish Centre for Expertise in Rheumatology at the Danish Hospital for Rheumatic Diseases, Department of Regional Health Research (IRS), University of Southern Denmark (SDU)
Locations (1):
- Danish Hospital for Rheumatic Diseases, Sønderborg, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No